CLINICAL TRIAL: NCT07145827
Title: Effect of Metformin on Endometrial Thickness in Postmenopausal Breast Cancer Patients Receiving Tamoxifen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uruk University (Other)
Responsible Party: Principal Investigator, Ghasak kais Abdulhussain, Lecturer in department of Pharmacology (B.Sc , M.Sc, Ph.D) / College of Pharmacy, Uruk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: UU-TAM-MET-2024-01
Record Dates: First submitted 2025-08-18; First posted 2025-08-28 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer; Endometrial Hyperplasia and Endometrial Cancers
Keywords: Metformin; Tamoxifen; Breast cancer; endometrial hyperplasia
MeSH Terms: conditions — Breast Neoplasms; Endometrial Hyperplasia; Endometrial Neoplasms | interventions — Tamoxifen

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: This is a double-blind study. Neither the participants nor the ultrasound operator assessing the primary outcome (endometrial thickness) will be aware of the treatment allocation. Study medication and placebo will be identical in appearance and packaging. Randomization codes will be securely held and only revealed after completion of data analysis, unless required for patient safety.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tamoxifen + Metformin (Experimental): Participants in this arm (n=30) will continue taking the standard oncological tamoxifen dose as prescribed and receive an addition of metformin 500mg twice daily, titrated to tolerance, during the 12-month study period.
  Interventions: Drug: Metfomin; Drug: tamoxifen
- Tamoxifen + Placebo (Placebo Comparator): Participants in this arm (n=30) will continue to receive the standard oncological dose of tamoxifen as prescribed, in addition to a placebo tablet matching the shape size and color of metformin tablet twice daily during the 12 months study period; they will act as the control group.
  Interventions: Drug: tamoxifen; Drug: Placebo matching Metformin

INTERVENTIONS:
Drug: Metfomin — Metformin Tab. 500mg twice daily for 12 months (titrated to tolerance if needed).
  Arms: Tamoxifen + Metformin
Drug: tamoxifen — Standard prescribed oncological dose.
Drug: Placebo matching Metformin — An inert, film-coated tablet identical in appearance and packaging to metformin 500 mg (same size, shape, color, coating, weight, and dosing schedule), manufactured without active ingredient using standard excipients (e.g., microcrystalline cellulose, starch/croscarmellose, povidone, magnesium stearate) and identical film coat (e.g., hypromellose, polyethylene glycol, titanium dioxide). Packaged in sealed blisters to minimize odor/taste cues. Dispensed by the investigational pharmacy per randomization; to be taken twice daily"
  Arms: Tamoxifen + Placebo

SUMMARY:
The goal of this clinical trial is to learn if metformin can reduce the increase in endometrial thickness caused by tamoxifen in women with estrogen-positive breast cancer taking tamoxifen for more than 1 year. It will also learn about the safety of taking metformin with tamoxifen. The main questions it aims to answer are:

1. Does metformin decrease endometrial thickness in women receiving tamoxifen?
2. What medical problems do participants have when taking metformin with tamoxifen?

Researchers will compare tamoxifen plus metformin to tamoxifen plus placebo to see if metformin works to reduce endometrial thickness compared to placebo patients.

Participants will:

1. Take metformin daily along with tamoxifen, or take tamoxifen with placebo.
2. Acquire baseline assessment and then visit the clinic at 3 months, 6 months, 9 months and 12 months for checkups and trans abdominal ultrasound test for endometrial thickness, and to be monitored for any side effects or complications.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal Female patients (amenorrhea ≥ 12 months).
* Histologically proven (Estrogen-positive) breast cancer.
* Completed all required surgery and/or chemotherapy (if indicated)
* On adjuvant tamoxifen for at least 1 year.
* Accepts to enroll in the study

Exclusion Criteria:

* Refusing to enroll in the study
* Ongoing or History of: endometrial or ovarian malignancy
* Concurrent hormonal therapy that might affect endometrial thickness
* Concurrent Diabetes mellitus in which metformin is prescribed.
* Known hypersensitivity or severe intolerance to metformin

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-01-02 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Change in endometrial thickness | Baseline, 3 months, 6 months, 9 months, and 12 months from enrollment
  Endometrial thickness will be measured using transabdominal ultrasound (in millimeters) by a trained radiologist. The primary outcome is the difference in endometrial thickness between the metformin plus tamoxifen group and the placebo plus tamoxifen control group.

CONTACTS AND LOCATIONS:
Overall Officials: Ghasak Kais Abdulhussain, BSc, MSc, PhD (Pharmacology), Principal Investigator — Uruk University
Locations (1):
- Baghdad Medical City / Department of Oncology, Baghdad, Baghdad Governorate, Iraq

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant-level data, including endometrial thickness measurements, baseline demographics, and follow-up data relevant to primary outcomes.
Time Frame: Upon publication of the trial result on open access repository.
Access Criteria: Access will be open to researchers and the public via a free, open-access data repository, with a DOI provided in the publication. Data will be de-identified to protect participant privacy.
URL: https://www.zenodo.org